CLINICAL TRIAL: NCT03891641
Title: A Momentum-enabled Treadling Methodology to Improve Gait and Enhance Mobility in Patients With Peripheral Arterial Disease
Brief Title: Momentum-enabled Treadling Methodology to Improve Gait and Enhance Mobility
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 continues to prevent recruitment of people over the age of 65 years.
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Treadwell Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-3169
Record Dates: First submitted 2019-03-25; First posted 2019-03-27 (Actual); Results first posted 2020-11-02 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-08

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized into a treadling group (n=15) or a control group (n=15). Treadling subjects will do so 3x per week (15 min sessions) for 6 weeks. The control group will be instructed to continue their normal daily activities.
Masking Description: No Masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treadling Group (Experimental): Treadling subjects will do so 3x per week (15 min sessions) for 6 weeks.
  Interventions: Behavioral: Treadwell Tredlr
- Control Group (No Intervention): Control Subjects continue their normal daily activities.

INTERVENTIONS:
Behavioral: Treadwell Tredlr — Complete treadling exercise 3x per week (15 min sessions) for 6 weeks.
  Arms: Treadling Group

SUMMARY:
This is a pilot study of a new exercise device (TREDLR) designed to facilitate repetitive ankle flexion/extension movements (i.e., "treadling") through a momentum-driven internal flywheel while seated. The specific goals of this project are to explore improvements in mobility and exercise capacity in individuals who treadle compared to a control group.

ELIGIBILITY:
Inclusion Criteria:

* Be able to walk without an assistive aid (i.e., walker, cane)
* Have the capacity the provide written informed consent
* Have previously diagnosed peripheral arterial disease (by self-report)

Exclusion Criteria:

* Lower extremity injury or fracture within the last 6 months
* Have a leg prosthesis
* Prisoners
* Individuals clearly lacking the capacity to provide informed consent
* Vestibular impairment

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Franz, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Applied Biomechanics Laboratory, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with the University of North Carolina.
Supporting Information: Study Protocol
Time Frame: Beginning 9 to 36 months following publication.
Access Criteria: The investigator who proposes to use the data must have approval from an IRB, IEC, or REB, as applicable, and execute a data use/sharing agreement with the University of North Carolina at Chapel Hill.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treadling Group | Control Group
Started | 10 | 7
Completed | 8 | 5
Not Completed | 2 | 2
Not completed — Study Stoppage Due to COVID-19 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treadling Group | Control Group | Total
Number analyzed (Participants) | 10 | 7 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 10 | 7 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.6 (5.4) | 71.3 (5.2) | 72.2 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 6 | 3 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 7 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 8 | 7 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 7 | 17

OUTCOME MEASURES:

1. Primary Outcome: Change in Overground Walking Speed After Intervention
Description: Measured from the time taken to walk 6 meters.
Time Frame: Baseline, 6 weeks
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Treadling Group | Control Group
Number analyzed (Participants) | 8 | 5
m/s | -0.046 (0.099) | 0.022 (0.140)

2. Primary Outcome: Change in 6-min Walk Distance
Description: Measured from the distance walked in 6 minutes.
Time Frame: Baseline, 6 weeks
Measure: Mean (Standard Deviation); unit: m
Arm/Group | Treadling Group | Control Group
Number analyzed (Participants) | 8 | 5
m | 13.60 (52.60) | 16.04 (38.40)

3. Secondary Outcome: Change in Stride Length
Description: Measured using motion capture as the distance between heel markers across successive steps.
Time Frame: Baseline, 6 weeks
Measure: Mean (Standard Deviation); unit: m
Arm/Group | Treadling Group | Control Group
Number analyzed (Participants) | 8 | 5
m | 0.005 (0.075) | -0.014 (0.016)

4. Secondary Outcome: Change in Peak Ankle Power
Description: Measured using motion capture and instrumented treadmill forces as the peak positive power generated by the calf muscles during the push-off phase of walking.
Time Frame: Baseline, 6 weeks
Measure: Mean (Standard Deviation); unit: W/kg
Arm/Group | Treadling Group | Control Group
Number analyzed (Participants) | 8 | 5
W/kg | -0.294 (0.630) | 0.088 (0.255)

ADVERSE EVENTS:
Time Frame: From the time of enrollment through the completion of the second laboratory session (i.e., post-test), approximately 6 weeks after the first laboratory session (i.e., baseline)
Arm/Group | Treadling Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/7
Other Adverse Events (participants affected / at risk) | 0/10 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-26): https://cdn.clinicaltrials.gov/large-docs/41/NCT03891641/Prot_SAP_000.pdf